CLINICAL TRIAL: NCT01280877
Title: Multicenter Study of Paraorbital-Occipital Alternating Current Stimulation Therapy in Patients With Optic Neuropathy
Brief Title: Paraorbital-Occipital Alternating Current Stimulation Therapy for Optic Neuropathy (MCT_optnerve)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Magdeburg (Other)
Collaborators: EBS Technologies GmbH (Industry)
Responsible Party: Principal Investigator, Bernhard A. Sabel, Principle PI, University of Magdeburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EBS-PP-2010-08-10-001
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Optic Nerve Diseases; Optic Nerve Injuries; Optic Neuropathies
Keywords: optic neuropathy; visual field; electric stimulation; alternating current; perimetry
MeSH Terms: conditions — Optic Nerve Diseases; Optic Nerve Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum stimulation (Experimental): Complete treatment with transorbital alternating current stimulation (tACS)
  Interventions: Device: tACS
- Sham stimulation (Sham Comparator): Same electrode montage set-up is used during tACS- and placebo-stimulation. Sham stimulation condition consists of minimal treatment with low intensity/few impulses tACS.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: tACS — Transorbital alternating current stimulation (tACS) is applied with a multi-channel device with paraorbital montage of 4 stimulation electrodes generating weak current pulses in predetermined firing bursts of 8 to 14 pulses. The amplitude of each current pulse was below 1000 microA. Current intensity was individually adjusted according to how well patients perceived phosphenes, i.e. any sensation of flickering light in response to the rtACS stimulation.
  Arms: Verum stimulation
Device: Sham stimulation — tACS is applied with the same device with equal electrodes set-up procedures but only one of four channels actually delivers current. The current intensity of this channel is individually adjusted (preselected on the side of lesioned eye) according with patient able to clearly perceive single phosphenes or any skin irritation phenomena (like weak sense of needles or vibration) whenever a single pulse is applied. The amplitude of pulses is always below 1000 microA. Current pulses are given as 1 pulse per minute during 25-35 min of session time. Session duration is equal for verum and sham patients. The perception of the single pulses leaves sham patients at the impression that they might receive the verum intervention, but total number of pulses is less than 0,5% of verum tACS.
  Arms: Sham stimulation

SUMMARY:
Aim is to validate that non-invasive brain stimulation can increase cortical excitability in the visual system. The investigators assess if transcranial alternating current stimulation (tACS) can improve visual field size in patients with optic nerve damage. Hypothesis: tACS would improve visual functions within the defective visual field (primary outcome measure).

DETAILED DESCRIPTION:
In addition, the correlation between the brain-derived neurotrophic factor (BDNF) or other plasticity markers are correlated to the improvement of the visual field after stimulation.

ELIGIBILITY:
Inclusion Criteria:

* patients with optic nerve lesion
* stable visual field defect with residual vision
* lesion age at least 6 months
* age at least 18 years
* no completely blindness, residual vision still existent

Exclusion Criteria:

* electric or electronic implants, e.g. heart pacemaker
* any metal artefacts in head and truncus
* epilepsy
* auto-immune diseases in acute stage
* mental diseases, e.g. schizophrenia etc.
* unstable diabetes, diabetes causing diabetic retinopathy
* addiction
* high blood pressure (max. 160/100 mmHg)
* instable or high level of intraocular pressure (i.e. > 27 mmHg)
* retinitis pigmentosa
* pathological nystagmus
* presence of an un-operated tumor anywhere in the body
* pregnant or breast-feeding women
* photo sensibility
* Fundus hypertonicus
* acute conjunctivitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Detection accuracy (DA) change in percent over baseline within defective visual field | Baseline - 8 weeks after stimulation; First follow-up 2 days after treatment course; Second follow-up 8 weeks after treatment course
  Central visual fields assessed with computer-based high-resolution perimetry (HRP). Based on such plots, areas of the visual field are characterized as intact, partially damaged or absolutely impaired (blind). Detection accuracy (DA) change in percent above baseline within defective visual field sectors is defined as the primary outcome criterion.

SECONDARY OUTCOMES:
DA change in percent over baseline regarding the damage region of the tested visual field (computer-based high-resolution perimetry) | Baseline - 8 weeks after stimulation; First follow-up 2 days after treatment course; Second follow-up 8 weeks after treatment course
  This parameter includes also intact sectors that are tested with HRP. It is hypothesized that improvements of the primary outcome criterion will outweigh the relative change in intact sectors as measured with HRP.
EEG parameters | Baseline - 8 weeks after stimulation; First follow-up 2 days after treatment course; Second follow-up 8 weeks after treatment course
  EEG power spectra
Reaction time change in ms | Baseline - 8 weeks after stimulation; First follow-up 2 days after treatment course; Second follow-up 8 weeks after treatment course
  Reaction time (RT) in HRP
Visual acuity (VA) | Baseline - 8 weeks after stimulation; First follow-up 2 days after treatment course; Second follow-up 8 weeks after treatment course
DA in static and kinetic conventional perimetry | Baseline - 8 weeks after stimulation; First follow-up 2 days after treatment course; Second follow-up 8 weeks after treatment course

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard A Sabel, Prof. Dr., Principal Investigator — Direktor, Institut für Medizinische Psychologie, Leipziger Str. 44, D-39120 Magdeburg, Germany
Locations (4):
- Germany (4):
  - Klinik für Neurologie, Charité Campus Mitte, Universitätsmedizin Berlin, Berlin
  - Klinische Neurophysiologie & Abteilung Augenheilkunde, Universitätsmedizin Göttingen, Göttingen
  - Augenklinik Kassel am Klinikum Kassel GmbH, Kassel
  - Inst. f. Medizinische Psychologie, Universitätsklinikum Magdeburg, Magdeburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gall C, Schmidt S, Schittkowski MP, Antal A, Ambrus GG, Paulus W, Dannhauer M, Michalik R, Mante A, Bola M, Lux A, Kropf S, Brandt SA, Sabel BA. Alternating Current Stimulation for Vision Restoration after Optic Nerve Damage: A Randomized Clinical Trial. PLoS One. 2016 Jun 29;11(6):e0156134. doi: 10.1371/journal.pone.0156134. eCollection 2016. PMID 27355577